CLINICAL TRIAL: NCT02436590
Title: A Prospective, Randomized, Double-Blind, Placebo Controlled Study to Evaluate Efficacy and Safety of an Active Pulsed Electromagnetic Field for the Treatment of Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of an Active Pulsed Electromagnetic Field for the Treatment of Osteoarthritis of the Knee
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-1403PSOA
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee; pulsed electromagnetic fields; PEMF
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active PEMF (Active Comparator): Subjects have a 2 out of 3 chance to get the active device which emits a Pulsed Electromagnetic Field (PEMF) from the Physio-Stim Model 3315OA device. Double blind randomization
  Interventions: Device: Orthofix Physio-Stim Model 3315OA
- Control/no PEMF (Placebo Comparator): Subjects have a 1 out of 3 chance of getting the control/placebo device which does not emit Pulsed Electromagnetic Field (PEMF) from the Physio-Stim Model 3315A device. Double blind randomization
  Interventions: Device: Orthofix Physio-Stim Model 3315OA

INTERVENTIONS:
Device: Orthofix Physio-Stim Model 3315OA — Active device emits PEMF signal; placebo/control device does not emit PEMF signal

SUMMARY:
The hypothesis of this study is that exposure to PEMF alters the cytokine environment of OA joints associated with a reduction of inflammation and improved homeostasis of the extracellular matrix (ECM), both potentially effecting symptomatic relief of OA pain, reducing cartilage breakdown, stimulate new cartilage formation therefore preserving joint structure.

DETAILED DESCRIPTION:
The hypothesis of this study is that exposure to PEMF alters the cytokine environment of OA joints associated with a reduction of inflammation and improved homeostasis of the extracellular matrix (ECM), both potentially effecting symptomatic relief of OA pain, reducing cartilage breakdown, stimulate new cartilage formation therefore preserving joint structure. The primary objective of this study is to prospectively determine, at 12 months post treatment, the safety and efficacy of treating OA of the knee with PEMF. Safety will be assessed through adverse event collection. Study subjects will be randomized in a 2:1 ratio (active: placebo control) to either an active or placebo control (inactive) Physio-Stim device. The study is powered to detect a significant difference between groups when 120 subjects (80 active: 40 placebo control) have completed the study. Planned enrollment for the study is 150 subjects, to allow for an attrition rate of 20%.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to wear the investigational device so that there is adequate PEMF exposure to the knee.
2. Subject must have a body mass index ≤ 45 at the time of consent.
3. Subject must be at least forty (≥ 40) years of age of age at the time of consent.
4. Subject must have an established diagnosis of primary femorotibial OA in the target knee by modified American College of Rheumatology criteria for at least 6 months and at least one of the following:

   i. Stiffness less than 30 min ii. Crepitus (noise or cracking on knee motion)
5. Subject must have symptomatic Kellgren-Lawrence (K-L) Grades 1-3 OA by radiograph (PA flexion) within 90 days of screening, where the K-L grades are defined as:

   Grade 1: doubtful narrowing of joint space and possible osteophytic lipping; Grade 2: definite osteophytes and definite narrowing of joint space; Grade 3: moderate multiple osteophytes and definite narrowing of joint space and some sclerosis and possible deformity of bone contour
6. Subject must have a visual analog pain score between 4 cm and 8 cm on a 10 cm scale in the target knee at the time of screening.
7. Subject must have a normal tibiofemoral angle (0-8°) and a joint space width of ≥ 3mm confirmed by radiograph.
8. Subject must be ambulatory.
9. Subject must NOT have had arthroscopy within 8 weeks of randomization.
10. Subject must NOT have had viscosupplementation within 8 weeks of randomization.
11. Subject must NOT have had NSAIDs within 1 week of randomization (low-dose aspirin as cardioprotective prophylaxis is permitted).
12. Subject must be willing to discontinue corticosteroids administered by any route except intranasal spray, steroid- containing ophthalmic solutions and anti-asthmatics.
13. Subject must be willing to take acetaminophen (up to 3000 mg/day) as pain medication for the duration of the study. Other pain medications may be allowed during the course of the study if the subject meets specific criteria.
14. Subject must be willing to STOP taking any pain medications 24 hours prior any scheduled study visit.
15. Subject must NOT have participated in a clinical study within the past 12 weeks that required the use of an investigational device, drug or biologic.
16. Subjects must be proficient in English.
17. Subject must be willing and able to sign an informed consent document.
18. Subjects must be willing and able to comply with all study procedures for the duration of the clinical study.

Exclusion criteria:

1. Subjects who have a body mass index > 45 at the time of consent.
2. Subjects with a diagnosis of inflammatory arthritis (rheumatoid arthritis, gout, joint infection, Lyme disease, SLE, etc.).
3. Subjects with a diagnosis of secondary arthritis (acromegaly, Charcot's arthropathy, hemochromatosis, Wilson's disease, ochronosis, etc.).
4. Subjects with confounding factors such as ipsilateral hip OA or chronic pain syndromes (fibromyalgia, Crohn's disease, ulcerative colitis, interstitial cystitis).
5. Subjects who have had an injury or an acute traumatic injury to the index knee within 6 months of screening will be excluded.
6. Subjects who have had treatment of the target knee with intra-articular injections of steroids within 8 weeks of screening.
7. Subjects who have had intra-articular injections of hyaluronic acid within 8 weeks of screening.
8. Subjects who plan to have surgery on the target knee within the study period.
9. Subjects who have used electrotherapy or acupuncture for OA of the target knee within 4 weeks of screening.
10. Subjects with significant and clinically evident mal-alignment of the target knee (> 10 degrees varus or valgus in the target knee).
11. Subjects with surgical metallic hardware in the target knee.
12. Subjects with pain in any other area of the lower extremities or back that is equal to or greater than the pain in the target knee.
13. Subjects who have contraindications to MRI and X-rays, for example, implanted electrical devices (cardiac pacemakers, deep brain stimulators).
14. Subjects with a current malignancy or who have received treatment for malignancy with the last 5 years, with the exception of resected basal cell carcinoma and squamous cell carcinoma of the skin.
15. Subjects who have an active substance abuse problem (drugs or alcohol) or a history of chronic substance abuse (> 5 years).
16. Subjects with skin breakdown or infection in the area where the study device will be placed.
17. Subjects with any chronic conditions (e.g., diabetes, hypertension, congestive heart failure, etc.) that have not been well-controlled for at least 3 months prior to screening.
18. Subjects who have any ongoing litigation for worker's compensation.
19. Subjects with any condition, in the opinion of the Investigator that might interfere with the evaluation of the study objectives.
20. Subjects who are unwilling or unable to adhere to the follow up schedule and procedures.
21. Subjects who are pregnant.
22. Subjects who are prisoners.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
change over time in WOMAC score | 6 mo, 12 mo
  The primary outcome variables are a statistically significant improvement in Western Ontario and McMaster Universities Arthritis Index (WOMAC) scores and by a significantly increased number of study subjects achieving minimally clinical important differences (MCIDs).

CONTACTS AND LOCATIONS:
Overall Officials: Roy K Aaron, MD, Principal Investigator — Warren Alpert Medical School of Medicine, Brown University, Providence, Rhode Island; Ronald Delanois, MD, Principal Investigator — Rubin Institute for Advance Orthopedics, Sinai Hospital of Baltimore
Locations (2):
- United States (2):
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Cleveland Clinic, Cleveland, Ohio